CLINICAL TRIAL: NCT02159625
Title: A Study of the Use of Abdominal Compression Elastic Support (ACES) for Hemodialysis Patients
Brief Title: Abdominal Compression Elastic Support (ACES)
Acronym: ACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Global Monitors, Inc. (Industry)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G120243/S001
Record Dates: First submitted 2014-05-30; First posted 2014-06-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Intradialytic Hypotension
Keywords: Abdominal Compression Elastic Support; Hemodialysis; hypotension; occurrence rate
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abdominal Compression Elastic Support (Experimental): To compress the abdomen at 15 mmHg for 3 hours during the course of hemodialysis treatment.
  Interventions: Device: Abdominal Compression Elastic Support

INTERVENTIONS:
Device: Abdominal Compression Elastic Support — The ACES will be used for HD patients who have had IDH episodes in the last month. For these patients, the ACES will impose a compression pressure of 15 mmHg to compress the abdominal section over the last three hours of the HD treatment. This action can increase venous return and hence cardiac output to improve the cardiovascular function of the patient. In this way, the IDH episode may be prevented or reduced in severity. This use is much less cumbersome over the use of IAB in dealing with PDOH. We perform this trial study to show the use ACES is more effective than the Trendelenburg maneuver or the infusion of isotonic saline, for example.
  Other Names: ACES

SUMMARY:
Hemodialysis (HD) patients with end stage renal disease (ESRD) experience higher rates of cardiovascular (CV) morbidity and mortality than do the general population and many populations with other chronic diseases. This exceptional risk is explained in part by known risk factors, such as diabetes, hypertension, and other uremia-related factors, including vascular calcification and stiffness, autonomic dysfunction, and a high burden of circulating inflammatory mediators. Recent studies suggest that blood pressure variability, especially intra-dialytic hypotension (IDH) is the most significant risk factor for these CV events. Studies have also shown that the use of IAB is capable of improving cardiovascular function for avoiding or minimizing the development of an orthostatic hypotensive episode (OHE) in patients with autonomic dysfunction, orthostatic hypotension (OH) in diabetes patients and children with orthostatic intolerance, and post-dialytic orthostatic hypotension (PDOH).

The investigators propose a study to examine the use of an abdominal compression elastic support (ACES) to prevent the development of IDH in patients who are known to be prone to these episodes. The ultimate goal is to facilitate more effective and safer dialysis therapy. The ACES has a configuration that is similar to a back-support work belt or an inflatable abdominal band (IAB). All of these devices are wrapped around to compress the abdomen at the waist.

DETAILED DESCRIPTION:
I. Study Design: Biomedical

1. Controls will be used. For the safety of ACES five healthy subjects will be used as controls to assess the safety and tolerability of the device. The regular HD treatments of each study patient will serve as their own control in assessing the effect of ACES use on their HD treatments. The control data are derived from the treatment logs of four to eight HD regular treatments taken by the patient.
2. The study design is an open trial.
3. No placebo is involved
4. This is a single center study to be done only at the Medical Center of University of Virginia (UVa).

II. Human Participants Ages: 18 or older Sex: Male and Female Race: All

Subjects or Patients:

1. 5 healthy subjects and 20 dialysis patients to complete protocol.
2. There could be a 50% drop out rate for the dialysis patients.
3. 30 (Up to 5 healthy subjects and Up to 35 dialysis patients) will be enrolled at all sites
4. All 30 subjects and patients will sign a consent form under this protocol.
5. The estimated time line for the study is 100% enrollment within 10 months III. Statistical Considerations

<!-- -->

1. Is stratification/randomization involved? No
2. What are the statistical considerations for the protocol? In analyzing the data, if the systolic blood pressure (SBP) of a given patient compared with the first blood pressure reading after initiating dialysis is larger than the threshold 20 mmHg (condition A) or the decrease in mean arterial pressure is larger than 10 mmHg and the development of hypotensive symptoms (condition B), this session (hour) will be identified as an IDH session (hour). The data may be divided into two groups (one under condition A and one under condition B) for further analysis on the impact of the conditions on the effectiveness of ACES.

   In our study design, the countermeasure implemented in each "control" session may be different. Our study can lead to an answer on whether the use of ACES is more effective in alleviating IDH than the "control" countermeasure.

   The researchers will only handle the quantitative data and the analysis of enumeration and quantitative data. To assure integrity in and correctness of data analysis, all data will be forwarded to a statistician who is not physically involved with the study for an independent evaluation.
3. Provide a justification for the sample size used in this protocol.

   A. On the safety issue: Due to the low compression pressure and no adverse effects seen in the use of IAB, we expect that the investigators should not see the development of any adverse effect in the current clinical trial. When the investigators carry out 40 ACES session in Phase II and show no adverse effect, then the likely hood for an adverse effect to develop will be at most 2.5%. Even if the occurrence frequency were at 25%, a sample size of 16 sessions will be more than adequate to demonstrate the safety hypothesis with a confidence better than 99% (i.e. P<0.01).

   B. On the reduction in occurrence frequency. The patients participated in the study will have at least 2 episodes in a month. It can add up to an occurrence frequency of 25%. This is to say that 20 out of the 80 control sessions will have IDH developed. If the occurrence frequency is reduced to 12.5% (i.e. 12 sessions with IDH out of the 80 ACES sessions), the data of 80 ACES session will be adequate to show a confidence level of 99% by the chi square test (P<0.01) that the use of ACES is effective in reducing the occurrence frequency. On the other hand, if the frequency estimated from the data of Phase II is reduced to 18% (instead of 12.5%), then the data of 80 ACES sessions in Phase II will yield a χ2 of about 2.0. With data of 80 more ACES sessions in Phase II, the value of χ2 for the same decrease in occurrence frequency may increase to 4 to indicate that the reduction in occurrence frequency has a confidence level of 95% (P<0.05).

   The above computation analysis has been expanded to examine how test size and the values of occurrence rate affect the value of χ2 and subsequently whether the occurrence rate is significantly reduced with the use of ACES. The investigators find that the three test sizes (80 tests mentioned here, 160 tests and 480 periods mentioned later) set for use in the protocol are adequate to carry out the statistical determination.

   Currently the investigators do not have a certain way to predict when IDH will develop. Thus, the investigators consider each HD session done on the same patient as independent.
4. The investigators have worked with a retired statistician in designing this protocol.

IV. Biomedical Research

1. Healthy subjects:

   In order to fulfill the study statistical requirements, up to five (5) healthy subjects will be tested for safety and tolerability of wearing ACES for 3 hours. Each healthy individual will then wear the ACES for three consecutive hours in a supine or seated position, except for use of the restroom if needed, and assess the measured parameters.

   If no major concerns are identified with this healthy population the use of ACES device will be offered for use in dialysis patients who have three or more episodes of IDH in the 4 weeks leading up to recruitment.
2. Dialysis Patients

   Hemodialysis patients at the University of Virginia Kidney Center have their hemodialysis done in a seated position (30° to 90°). The investigators will be using the ACES device on these patients in a seated position.

   In order to fulfill the study statistical requirements, up to ten (10) ESRD patients on HD will be tested for safety and tolerability of wearing ACES during their dialysis sessions.

   Screening trial session for Dialysis Patients After the patient reads and signs the consent form and passes the inclusion and exclusion criteria, the investigators will have him or her to undergo a trial session of ACES. This trial session can be done on the same day as the consent form or it can be done on another day that the patient is coming for a regular dialysis session. This trial session is designed to find out whether the patient can tolerate the compression of the ACES and whether his/her SBP and heart rate can be significantly altered by the compression. Over the course of this screening trial, the patient will be advised that he can request removal of the ACES whenever he/she wishes.
3. Control & ACES Sessions:

   The patients will undergo a HD treatment as prescribed by their attending nephrologists. The investigators expect that the characteristics of these treatments will have the following general features:

   • The HD setting can lead to a Kt/V larger than 1.2

   • A procedure or countermeasure will have been prescribed and set up as standard of care to deal with the development of IDH.
   * The measurement of blood pressure and heart rate will be performed by the usual dialysis machine for a given patient, providing internal equipment standardization
   * The blood pressure cuff will be applied to bare skin on the patient's arm
   * The data obtained for eight regular HD treatments without wearing the ACES will be identified as the control data. For each patient, four HD treatment sessions will be conducted with the use of ACES in Phase II and four more will be done in Phase III if the data of Phase II calls for.

   Preparation to start the hemodialysis with ACES

   • Before the screening test of the patient, the investigators will get the waist circumference of the patient. The size of the ACES is chosen from this specification: 22"~27" (56~68cm)-Small, 28"~33" (71~84cm)-Medium, 34"~40" (86~101cm)-Large, 41"~47" (104~119cm)-Extra-Large, 48"~54" (122~137cm)-Extra-Extra-Large 55"~61" (140~155cm).

   • Put on the ACES with its band tips already aligned with the white marking. At this "no load" marking, the compression pressure imposed by the ACES is less than 2 mmHg. This step is done before the patient is seated and attached to the blood lines.

   • The HD treatment will start as usual.

   During HD Control and ACES session if the patient experiences IDH or SBP drop If the study investigators deem that the patient is experiencing symptoms of IDH or sees that the SBP drops 20 mm Hg, then a charted course will be used on what countermeasures are to be employed.

   Post-dialytic care and data collection • Post dialytic procedure and care will include:

   o Removal of the ACES and one more BP and pulse measurement,

   o Discharge of the patient who is diagnosed as having no PDOH,

   o Whether the patient is asked to come back for another HD treatment the next day,

   o If the patient is classified as one with PDOH, the procedure to discharge the patient as prescribed by the physician will be followed. If it is prescribed to take a standing up test, it will be done with the ACES on. If the patient is to be sent home, then the ACES will be taken off the patient and another standing up test be done. If the patient is to be sent to an emergency center, then the physician will make a decision on whether to send the patient with the ACES on or with it off.
4. Events calling for decompression of the ACES.

If the following complications develop while the ACES is in use the device will be removed • A decrease in toe O2 saturation below 90%, • An increase in leg circumference by more than 10% to indicate leg edema,

• Pain or cramping in the abdominal area and/or lower extremities being more severe than the norm

* Vomiting more severe than the norm
* Any other threatening complication
* The patient requests removal of the device (reason for request will be recorded)

The study team will investigate whether the complications result from abdominal compression imposed by the ACES. If ACES is deemed as the cause, then the ACES will be decompressed. When the level of aspartate aminotransferase (AST) alanine aminotransferase (ALT) become available to Global Monitor, Inc. and is found to be higher than the norm, then a retrospective analysis will be made to determine whether the level increase relates to the use of ACES.

V. Data and Safety Monitoring Plan An adverse event will be considered any undesirable sign, symptom or medical or psychological condition even if the event is not considered to be related to the investigational drug/device/intervention. Medical condition/diseases present before starting the investigational drug/intervention will be considered adverse events only if they worsen after starting study treatment/intervention. An adverse event is also any undesirable and unintended effect of research occurring in human patients as a result of the collection of identifiable private information under the research. Adverse events also include any problems associated with the use of an investigational device that adversely affects the rights, safety or welfare of patients.

The symptoms or disease developments described as the exclusion criteria (i.e. beyond the first six) will be considered as adverse effect. The symptoms or excessive decrease in SBP, for example, that are normally associated with hypotension development and are found to be common in HD patients of UVa clinics will be reported but not considered as adverse event and not used as a trigger to discontinue the ACES session.

The adverse event will be reported to FDA in a case report form.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to give informed consent for participation in this study
* Age ≥ 18 years
* A body weight > 100 lb or a body mass index > 18.5.
* End-stage renal disease with hemodialysis in-center three times per week
* Not missing any treatments in the preceding two weeks and in compliance with instructions from the health care provider.
* In the last month had at least two episodes of IDH (defined as having hypotensive symptoms such as dizziness, fainting, headache, nausea, vomiting, cramping, weakness, blurry vision and/or a decrease in systolic blood pressure (SBP) of more than 20 mmHg).
* Hemoglobin greater than or equal to 9.0 g/dL (hematocrit 27%) to hemoglobin of 15.0 g/dL (hematocrit 45%).

Exclusion Criteria:

* • Pregnancy (self-reported)
* Allergic to nylon, polyesters and latex.
* Not able to understand the English language
* Not able to disengage the ACES from compression
* Having an excessively low systolic blood pressure (SBP which is less than 90 mmHg)
* Hemoglobin less than 9.0 g/dL or greater than 15 g/dL
* Excessive intra-abdominal fluid pressure
* Respiratory distress
* Bleeding in the chest and abdomen
* Bleeding dyscrasia causing serious coagulation problem
* Raised intra-abdominal pressure
* Having the following cardiovascular, pulmonary and abdominal complications:

  * Systolic congestive heart failure, defined as a systolic ejection fraction of less than 25%
  * Coronary artery disease defined as having a history of myocardial infarction or hemo-dynamically significant stenosis on cardiac catheterization or acute or chronic angina
  * Circulatory shock
  * Head trauma and/or abdominal trauma in the past three months
  * Mesenteric ischemia
  * Active foot ulcer
  * Pulmonary edema
  * Uncontrolled Hypertension (defined as systolic pressure of 180 mm Hg or a diastolic pressure of 110 mm Hg or higher) - using the average blood pressures obtained at one prior recent dialysis session and the average blood pressures obtained at the screening trial session for ACES.
  * Liver disease as defined as an elevated ALT, AST, and Alkaline Phosphatase 2.5 times the upper limit of normal on a prior lab from medical records.
  * INR > 1.5 or use of coumadin
  * Platelets < 100
  * Active infection
  * The need to use anti-hypotensive drugs on the days the ACES belt is applied.
  * If the average systolic blood pressure with anti-hypotensive drugs or without and made before hemodialysis treatment is less than 90 mmHg, then the ACES session will be postponed to the next treatment. If similar hypotension situation occurs in the next ACES/hemodialysis treatment, then the subject will be taken out of the ACES trial and be considered a screen fail.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The number of HD sessions or hourly periods of the sessions being classified as IDH episode, which indicates that the patient's SBP decreases more than 20 mmHg from the SBP at the start of HD session or the patient experiences hypotensive symptoms. | 4 hours of each HD session
  This is an efficacy measure of the use of ACES to alleviate IDH. The investigators count the number of sessions with IDH and non-IDH sessions for the control ones and ACES sessions and use the Chi-square analysis to answer whether there is a significant reduction in the occurrence frequency of IDH. The investigators will examine in a similar way the counts based on the IDH development in the four hourly periods within a HD treatment for controls and those with ACES.

SECONDARY OUTCOMES:
The change in ALT and AST over the course of HD sessions with ACES | 4 hours for each HD session
  One blood sample is taken before the start of the HD session and the other at the end of the session. The investigators then measure the ALT and AST level of the samples. A student paired t-test will be used to examine whether the use of ACES increases the level of ALT and AST. If the result indicates insignificant increase, the investigators can then conclude that the use of ACES imposes no damage to the liver.

OTHER OUTCOMES:
Dry weight, pre- and post-dialysis weight (kg) of the control and ACES HD sessions. | 4 hours
  A student paired t-test will be used to examine whether the use of ACES alters the these weights beyond the control ones.
The achieved UF in comparison with the ultrafiltration (UF) goal set by the physician. | 4 hours
  This is an assessment on the effectiveness of HD process and on whether it is affected with the use of ACES. A student paired t-test will be used.
Number and type of countermeasures employed to counter the IDH development in control and ACES sessions. | 4 hours
  This is an assessment on the effectiveness of ACES on whether it reduces the need to call for additional countermeasures. A student t-test will be used to analyze the number data.
Prescribed and delivered time of the HD session. | 4 hours
  This is an assessment on the effectiveness of HD process and on whether it is affected with the use of ACES. On the latter, a student paired t-test will be used to compare the difference between prescribed and delivered time to find out whether the difference is altered for the ACES session.
Achieved Kt/V | 4 hours
  This is an assessment on the effectiveness of HD process and on whether the set Kt/V is achieved for ACES sessions. A student paired t-test will be used.
Recovery time after HD session | at 4 hours after the HD session
  The recovery time will be considered as a quality assessment of the HD treatment. By a student paired t-test, we may find out whether the use of ACES will lead to faster recovery for the patients.
Record of patient's tolerance to the use of ACES, comments on discomfort associated with HD process, and likelihood to use ACES for future HD treatments. | 4 hours
  These parameters, in the form of yes or no, are subjectively provided by the patient for the investigators to assess whether the ACES will induce discomfort to the patient taking HD and whether they want to use ACES again.

CONTACTS AND LOCATIONS:
Overall Officials: Kline Bolton, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Coll E, Valles M, Torguet P, Bronsoms J, Mate G, Mauri JM. [Evaluation of plasma volume variation during different hemodialysis maneuvers]. Nefrologia. 2004;24(5):463-9. Spanish. PMID 15648904
- [Background] Dheenan S, Henrich WL. Preventing dialysis hypotension: a comparison of usual protective maneuvers. Kidney Int. 2001 Mar;59(3):1175-81. doi: 10.1046/j.1523-1755.2001.0590031175.x. PMID 11231376
- [Background] Lee JS. 1998 Distinguished Lecture: biomechanics of the microcirculation, an integrative and therapeutic perspective. Ann Biomed Eng. 2000 Jan;28(1):1-13. doi: 10.1114/1.249. PMID 10645783
- [Background] Lindsay RM, Heidenheim PA, Nesrallah G, Garg AX, Suri R; Daily Hemodialysis Study Group London Health Sciences Centre. Minutes to recovery after a hemodialysis session: a simple health-related quality of life question that is reliable, valid, and sensitive to change. Clin J Am Soc Nephrol. 2006 Sep;1(5):952-9. doi: 10.2215/CJN.00040106. Epub 2006 Jul 6. PMID 17699312
- [Background] Smit AA, Wieling W, Fujimura J, Denq JC, Opfer-Gehrking TL, Akarriou M, Karemaker JM, Low PA. Use of lower abdominal compression to combat orthostatic hypotension in patients with autonomic dysfunction. Clin Auton Res. 2004 Jun;14(3):167-75. doi: 10.1007/s10286-004-0187-x. PMID 15241645
- [Background] Tanaka H, Yamaguchi H, Tamai H. Treatment of orthostatic intolerance with inflatable abdominal band. Lancet. 1997 Jan 18;349(9046):175. doi: 10.1016/S0140-6736(97)24003-1. No abstract available. PMID 9111544
- [Background] Yamamoto N, Sasaki E, Goda K, Nagata K, Tanaka H, Terasaki J, Yasuda H, Imagawa A, Hanafusa T. Treatment of post-dialytic orthostatic hypotension with an inflatable abdominal band in hemodialysis patients. Kidney Int. 2006 Nov;70(10):1793-800. doi: 10.1038/sj.ki.5001852. Epub 2006 Sep 27. PMID 17003821
- [Background] Palmer BF, Henrich WL. Recent advances in the prevention and management of intradialytic hypotension. J Am Soc Nephrol. 2008 Jan;19(1):8-11. doi: 10.1681/ASN.2007091006. PMID 18178796
- [Background] Lee, JS, Current Status on Countermeasures for Intradialytic Hypotension, in "Tributes to Yuan-Cheng Fung on His 90th Birthday, Biomechanics, from Molecules to Man", ed. S. Chien et al, World Scientific, Singapore, 219-230, 2010.
- [Background] Lee, JS, The Role of Microcirculation in Intradialytic Hypotension. Dialysis Times, 18:3-4, 2011
- [Background] Denq JC, Opfer-Gehrking TL, Giuliani M, Felten J, Convertino VA, Low PA. Efficacy of compression of different capacitance beds in the amelioration of orthostatic hypotension. Clin Auton Res. 1997 Dec;7(6):321-6. doi: 10.1007/BF02267725. PMID 9430805